CLINICAL TRIAL: NCT05436171
Title: Prevalence of Obstetric Anal Sphincter Injury With a Reducing Episiotomy Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LAU Yan Yan, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE 2022.259
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Anal Sphincter Injury
Keywords: Anal sphincter injury; Episiotomy; Prevalence; OASIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All deliveries conducted from 2011 to 2021 in Prince of Wales Hospital: All deliveries conducted from 2011 to 2021 in Prince of Wales Hospital
  The target sample size will be about 67,000 women who had delivered in our unit from 2011 to 2021. Among them, it is expected that 75-80% had vaginal deliveries, either normal vaginal delivery or instrumental delivery. 53,600 will be recruited in study site.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Obstetric anal sphincter injury (OASIS) is a serious complication of a vaginal delivery. High proportion of women, 40-59%, suffer from faecal incontinence (FI) after this type of injury.1-3 OASIS and FI have a negative impact on women's quality of life.4 The rate of elective caesarean section at second birth was much higher in women with OASIS at first birth compared with women without the injury (adjusted odds ratio 18.3, 95% CI 16.4-20.4).5 Primiparity has an increased risk of OASIS (odds ratio (OR) 2.39-8.34).6,7 Other factors are macrosomia and instrumental vaginal delivery.6,7 The role of episiotomy on OASIS has also been widely studied but there are controversial results.

There were around 500-7000 deliveries at Prince of Wales Hospital annually. Among them, 50-55% was nulliparous women. About 65 -70% of women had normal vaginal delivery and another 5-10% had instrumental delivery. There was a change from 'routine episiotomy' to a more restrictive use of episiotomy in normal vaginal delivery during the last 10 years, with a reduction of rate of episiotomy from 90% to about 50% (from Dept.'s internal audit). The objective of this study is to evaluate the prevalence of OASIS in the era of a reduction of episiotomy.

DETAILED DESCRIPTION:
Obstetric anal sphincter injury (OASIS) is a serious complication of a vaginal delivery. High proportion of women, 40-59%, suffer from faecal incontinence (FI) after this type of injury.1-3 OASIS and FI have a negative impact on women's quality of life.4 The rate of elective caesarean section at second birth was much higher in women with OASIS at first birth compared with women without the injury (adjusted odds ratio 18.3, 95% CI 16.4-20.4).5 Primiparity has an increased risk of OASIS (odds ratio (OR) 2.39-8.34).6,7 Other factors are macrosomia and instrumental vaginal delivery.6,7 The role of episiotomy on OASIS has also been widely studied but there are controversial results.

Episiotomy is a surgical enlargement of the vaginal orifice by an incision to the perineum during the last part of the second stage of labour or delivery.8 It is accepted that episiotomy facilitates delivery, prevents perineal lacerations and undue stretching of the pelvic floor.9 It is also believed that an episiotomy is easier to repair and heals better than a tear.10 Mediolateral episiotomy is the most frequently used type of episiotomy in Hong Kong. Some obstetric units perform episiotomy more liberally on a routine basis; while others adopt a more restrictive policy. Cochrane review identified eight randomized controlled trials (RCT) comparing routine episiotomy and restrictive episiotomy. 9,10-17 The restrictive use of episiotomy shows a lower risk of severe perineal trauma (relative risk (RR) 0.67, 95% CI 0.49-0.91), posterior perineal trauma (RR 0.88, 95% CI 0.84-0.92), need for suturing perineal trauma (RR 0.71, 95% CI 0.61-0.81), and healing complications at seven days (RR 0.69, 95% CI 0.56-0.85).13 No difference is shown in the incidence of major outcomes such as severe vaginal and perineal trauma (when both vaginal and perineal trauma are counted) nor in pain, dyspareunia or urinary incontinence. However, the restrictive use of episiotomy has an increased risk of anterior perineal trauma (RR 1.84, 95% CI 1.61-2.10).13 Therefore, it is not advised to practice routine episiotomy.

From a large retrospective studies conducted in Caucasian countries, mediolateral episiotomy has been shown to protect women from OASIS (OR 0.21-0.54). 6,7,18 Besides, there was also evidence showing that Asian women delivered in Caucasian countries with a low episiotomy rate had a high risk of OASIS.19,20 Furthermore, ethnical difference in pelvic connective tissues have been reported.21 And pregnant Chinese women has been shown to smaller genital hiatus and less mobility of pelvic organs than pregnant Caucasian women.22 This may lead to a different outcome in perineal trauma in Asian women with or without episiotomy during vaginal delivery.

There were around 500-7000 deliveries at Prince of Wales Hospital annually. Among them, 50-55% was nulliparous women. About 65-70% of women had normal vaginal delivery and another 5-10% had instrumental delivery. There was a change from 'routine episiotomy' to a more restrictive use of episiotomy in normal vaginal delivery during the last 10 years, with a reduction of rate of episiotomy from 90% to about 50% (from Dept.'s internal audit). The objective of this study is to evaluate the prevalence of OASIS in the era of a reduction of episiotomy. This would help inform obstetricians and midwives if there is any change in rate of OASIS and the relationship with episiotomy. The information would be useful to counsel our patients.

The protocol of current study complies with Declaration of Helsinki.

The HA CMS OBSCIS is the electronic system that have collected the demographic, pregnancy, delivery and postnatal data of pregnant women. The data was entered by midwives and obstetricians during all consultations and admission of delivery of all pregnant women.

In this study, the following information will be retrieved from the CMS OBSCIS database for all delivery conducted from 2011 to 2021.

1. Demographic data: age, parity, body weight and height
2. Past obstetric history (if any): mode of delivery, birthweight and sex of infant, use of episiotomy
3. Delivery data: gestation at delivery, need of induction of labour, analgesics during labour, duration of labour, mode of delivery, use of episiotomy, any perineal tear, blood loss during delivery, need of transfusion, wound complication, duration of hospital stay; and infant's birthweight, sex and apgar score
4. For women with OASIS: the method of repair, the symptom of pelvic floor disorders, such as faecal or flatal incontinence, urinary incontinence, symptoms of prolapse after the delivery.

ELIGIBILITY:
Inclusion Criteria:

* All deliveries conducted from 2011 to 2021 in Prince of Wales Hospital

Exclusion Criteria:

* Deliveries with Caesarean Section

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who had delivered in our unit from 2011 to 2021
Study Population: The target sample size will be about 67,000 women who had delivered in our unit from 2011 to 2021. Among them, it is expected that 75-80% had vaginal deliveries, either normal vaginal delivery or instrumental delivery. 53,600 will be recruited in study site.
Sampling Method: Probability Sample
Enrollment: 6700 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of obstetric anal sphincter injury (third or fourth degree tear) detected clinically immediately after delivery | Immediately after delivery
  Prevalence of obstetric anal sphincter injury (third or fourth degree tear) detected clinically immediately after delivery

SECONDARY OUTCOMES:
The factors associated with OASIS | Immediately after delivery
  Linear regression will be used to assess the correlations between factors e.g. mode of delivery, episiotomy, perineal/vaginal tear, duration of labour, birthweight and OASIS. Univariate and multivariate analysis will be used to look for potential factors of OASIS.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yan Lau, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Norderval S, Nsubuga D, Bjelke C, Frasunek J, Myklebust I, Vonen B. Anal incontinence after obstetric sphincter tears: incidence in a Norwegian county. Acta Obstet Gynecol Scand. 2004 Oct;83(10):989-94. doi: 10.1111/j.0001-6349.2004.00647.x. PMID 15453900
- [Background] Sultan AH, Kamm MA, Hudson CN, Bartram CI. Third degree obstetric anal sphincter tears: risk factors and outcome of primary repair. BMJ. 1994 Apr 2;308(6933):887-91. doi: 10.1136/bmj.308.6933.887. PMID 8173367
- [Background] Sangalli MR, Floris L, Faltin D, Weil A. Anal incontinence in women with third or fourth degree perineal tears and subsequent vaginal deliveries. Aust N Z J Obstet Gynaecol. 2000 Aug;40(3):244-8. doi: 10.1111/j.1479-828x.2000.tb03330.x. PMID 11065029
- [Background] Tucker J, Clifton V, Wilson A. Teetering near the edge; women's experiences of anal incontinence following obstetric anal sphincter injury: an interpretive phenomenological research study. Aust N Z J Obstet Gynaecol. 2014 Aug;54(4):377-81. doi: 10.1111/ajo.12230. PMID 25117190
- [Background] Edozien LC, Gurol-Urganci I, Cromwell DA, Adams EJ, Richmond DH, Mahmood TA, van der Meulen JH. Impact of third- and fourth-degree perineal tears at first birth on subsequent pregnancy outcomes: a cohort study. BJOG. 2014 Dec;121(13):1695-703. doi: 10.1111/1471-0528.12886. Epub 2014 Jul 9. PMID 25040835
- [Background] de Leeuw JW, Struijk PC, Vierhout ME, Wallenburg HC. Risk factors for third degree perineal ruptures during delivery. BJOG. 2001 Apr;108(4):383-7. doi: 10.1111/j.1471-0528.2001.00090.x. PMID 11305545
- [Background] Aukee P, Sundstrom H, Kairaluoma MV. The role of mediolateral episiotomy during labour: analysis of risk factors for obstetric anal sphincter tears. Acta Obstet Gynecol Scand. 2006;85(7):856-60. doi: 10.1080/00016340500408283. PMID 16817086
- [Background] Thacker SB, Banta HD. Benefits and risks of episiotomy: an interpretative review of the English language literature, 1860-1980. Obstet Gynecol Surv. 1983 Jun;38(6):322-38. PMID 6346168
- [Background] Harrison RF, Brennan M, North PM, Reed JV, Wickham EA. Is routine episiotomy necessary? Br Med J (Clin Res Ed). 1984 Jun 30;288(6435):1971-5. doi: 10.1136/bmj.288.6435.1971. PMID 6428627
- [Background] House MJ, Cario G, Jones MH. Episiotomy and the perineum: a random controlled trial. J Obstet Gynaecol 1986;7:107-110
- [Background] Klein MC, Gauthier RJ, Jorgensen SH, Robbins JM, Kaczorowski J, Johnson B, Corriveau M, Westreich R, Waghorn K, Gelfand MM, et al. Does episiotomy prevent perineal trauma and pelvic floor relaxation? Online J Curr Clin Trials. 1992 Jul 1;Doc No 10:[6019 words; 65 paragraphs]. doi: 10.1097/00006254-199404000-00008. PMID 1343606
- [Background] Rodriguez A, Arenas EA, Osorio AL, Mendez O, Zuleta JJ. Selective vs routine midline episiotomy for the prevention of third- or fourth-degree lacerations in nulliparous women. Am J Obstet Gynecol. 2008 Mar;198(3):285.e1-4. doi: 10.1016/j.ajog.2007.11.007. Epub 2008 Jan 25. PMID 18221925
- [Background] Carroli G, Mignini L. Episiotomy for vaginal birth. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD000081. doi: 10.1002/14651858.CD000081.pub2. PMID 19160176
- [Background] Routine vs selective episiotomy: a randomised controlled trial. Argentine Episiotomy Trial Collaborative Group. Lancet. 1993 Dec 18-25;342(8886-8887):1517-8. PMID 7902901
- [Background] Dannecker C, Hillemanns P, Strauss A, Hasbargen U, Hepp H, Anthuber C. Episiotomy and perineal tears presumed to be imminent: randomized controlled trial. Acta Obstet Gynecol Scand. 2004 Apr;83(4):364-8. doi: 10.1111/j.0001-6349.2004.00366.x. PMID 15005784
- [Background] Eltorkey MM, Al Nuaim MA, Kurdi AM, Sabagh TO, Clarke F. Episiotomy, elective or selective: a report of a random allocation trial. Journal of Obstetrics and Gynaecology 1994;14:317-320.
- [Background] Sleep J, Grant A, Garcia J, Elbourne D, Spencer J, Chalmers I. West Berkshire perineal management trial. Br Med J (Clin Res Ed). 1984 Sep 8;289(6445):587-90. doi: 10.1136/bmj.289.6445.587. PMID 6432201
- [Background] Hauck YL, Lewis L, Nathan EA, White C, Doherty DA. Risk factors for severe perineal trauma during vaginal childbirth: a Western Australian retrospective cohort study. Women Birth. 2015 Mar;28(1):16-20. doi: 10.1016/j.wombi.2014.10.007. Epub 2014 Dec 1. PMID 25476878
- [Background] Grobman WA, Bailit JL, Rice MM, Wapner RJ, Reddy UM, Varner MW, Thorp JM Jr, Leveno KJ, Caritis SN, Iams JD, Tita ATN, Saade G, Rouse DJ, Blackwell SC, Tolosa JE, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Racial and ethnic disparities in maternal morbidity and obstetric care. Obstet Gynecol. 2015 Jun;125(6):1460-1467. doi: 10.1097/AOG.0000000000000735. PMID 26000518
- [Background] Davies-Tuck M, Biro MA, Mockler J, Stewart L, Wallace EM, East C. Maternal Asian ethnicity and the risk of anal sphincter injury. Acta Obstet Gynecol Scand. 2015 Mar;94(3):308-15. doi: 10.1111/aogs.12557. Epub 2015 Jan 10. PMID 25494593
- [Background] Zacharin R. "A Chinese anatomy" - the pelvic supporting tissues of the Chinese and Occidental female compared and contrasted. Aust N Z J Obstet Gynaecol 1977;17:1-11.
- [Background] Cheung RY, Shek KL, Chan SS, Chung TK, Dietz HP. Pelvic floor muscle biometry and pelvic organ mobility in East Asian and Caucasian nulliparae. Ultrasound Obstet Gynecol. 2015 May;45(5):599-604. doi: 10.1002/uog.14656. Epub 2015 Apr 6. PMID 25175901